CLINICAL TRIAL: NCT00658242
Title: Craniofacial Surgery Perioperative Registry
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Children's Anesthesiology Associates, Ltd. (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-3-5842
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Craniotomy
Keywords: craniofacial; maxillofacial; osteotomy; craniectomy; craniotomy

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- I: Subjects having Craniofacial surgery

SUMMARY:
Craniofacial reconstruction procedures are undertaken in young children to improve appearance, prevent functional disturbances, and enhance psychosocial development. These procedures involve wide scalp dissections and multiple osteotomies and have been associated with significant morbidity. The most commonly seen perioperative complications are associated with the rate and extent of blood loss. This prospective observational registry will be a research tool which will provide a means to evaluate perioperative management of these children at CHOP.

DETAILED DESCRIPTION:
Craniofacial reconstructive surgery involves a surgical approach to the craniofacial region to repair cranial vault and facial deformities. These procedures are undertaken in young children to improve appearance, prevent functional disturbances, and enhance psychosocial development. The surgery is extensive, often requiring wide scalp dissections and multiple osteotomies and has been associated with significant morbidity. Reported complications include intra-operative cardiac arrest, massive blood loss, intraoperative tracheal extubation, venous air embolism, hypotension, coagulopathy, bradycardia, postoperative seizures, surgical site infections, facial swelling, and unplanned postoperative mechanical ventilation. The most severe and commonly seen problems are associated with the rate and extent of blood loss. Studies report estimated blood loss to average between 60% and 100% of the patient's estimated blood volume, with a range of 20-500%.(Hildebrandt et al 2007) The accurate and timely estimation of blood loss is very difficult and results in imprecise quantitative and qualitative replacement. Clinically important hypotension, metabolic acidosis, anemia, polycythemia, dilutional coagulopathy, cardiac arrest, and death are all related to blood loss. The creation of this prospective observational registry will provide a means to describe the incidence of these and other clinically important perioperative problems.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females with ages from birth to 18 years.
2. Patients undergoing surgical procedures on the craniofacial region performed by plastic surgeons, neurosurgeons, or by plastic surgeons in concert with neurosurgeons.
3. Patients undergoing plastic surgical procedures involving a craniotomy, craniectomy, maxillofacial osteotomy, strip craniectomy, or other plastic surgical procedure involving bones of the head and face.
4. Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria:

1. Patients undergoing craniofacial plastic surgical procedures not involving bones of the head and face.
2. Patients not admitted to the intensive care unit following surgery.
3. Patients undergoing procedures only involving the mandible.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects presenting for craniofacial surgery
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2008-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To create a research tool that prospectively captures perioperative data in the craniofacial surgical patient population that may provide insights into the perioperative management and help guide clinical decision making. | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Stricker, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital Of Philadelphia, Philadelphia, Pennsylvania, United States